CLINICAL TRIAL: NCT05295914
Title: Performance of Novel Simplified Score for Chronic Hepatitis B Treatment Eligibility in Thailand
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Watcharasak Chotiyaputta, Associate professor, Faculty of Medicine, Siriraj Hospital, Mahidol University
Other Study IDs: Si 745/2021
Record Dates: First submitted 2022-03-07; First posted 2022-03-25 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Chronic Hepatitis B
Keywords: chronic hepatitis B, TREAT-B, REACH-B, WHO criteria
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with chronic hepatitis B infection: Patient with chronic hepatitis B infection visited at liver and internal medicine clinic, Siriraj hospital between January 2015-2020
  Interventions: Diagnostic Test: TREAT-B score

INTERVENTIONS:
Diagnostic Test: TREAT-B score — TREAT-B score: ALT(alanine transferase), HBeAg REACH-B score: sex, ALT, HBV viral load, age WHO-simplified score: ALT, cirrhosis
  Other Names: WHO simplified score; REACH-B score

SUMMARY:
International and national guideline for chronic hepatitis B (HBV) infection treatment recommend initiated antiviral in high HBV viral loads patients with significant liver inflammation and significant liver fibrosis. In Thailand, HBV viral loads and liver elastography are limited available in seconds to tertiary care hospital.

Recently, many of simplified scoring system (TREAT-B score, WHO (World Health Organization)-simplified score and REACH-B score) were developed for assessment of antiviral initiation.

This study aim to evaluate the performance of simplified score for chronic HBV treatment compare to Thailand and international standard guideline.

DETAILED DESCRIPTION:
According to WHO Global health sector strategy on viral hepatitis 2016- 2021, WHO aim to global eliminate HBV infection within 2030. Main strategies for achievement are effective prevention and treatment.

International and national guideline for HBV infection treatment recommend initiated antiviral in high HBV viral loads patients with significant liver inflammation and significant liver fibrosis. Thus, HBV viral load and liver elastography are required for indication assessment. In low-to-middle income country such as Thailand, HBV viral loads and liver elastography are limited available in seconds to tertiary care hospital.

Recently, many of simplified scoring system (TREAT-B score, WHO-simplified score and REACH-B score) were developed for assessment of antiviral initiation.

This study aim to evaluate the performance of simplified score for chronic HBV treatment compare to Thailand and international standard guideline.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naive chronic hepatitis B infection patients who visited at liver clinic and internal medicine clinic Siriraj hospital during January 2015-December 2021
* Age > 18 years

Exclusion Criteria:

* Treatment experience chronic hepatitis B infection patients
* HIV co-infection
* HCV (hepatitis C) co-infection
* concomitant HCC (hepatocellular carcinoma)
* Pregnancy
* Incomplete data

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Treatment naive chronic hepatitis B infection patients who visited at liver clinic and internal medicine clinic Siriraj hospital during January 2015-December 2021
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-04-10 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Performance of TREAT-B score for eligible antiviral treatment | at 1st OPD(out patient department) visit through initiation of antivirus or 1 year (if not indication for antivirus)
  Gold standard: Eligible antiviral treatment according to EASL (European Association for the Study of the Liver) criteria Description: performance was define by sensitivity(%), specificity(%), PPV(positive predictive value)(%), NPV (negative predictive value)(%), positive LR(likelihood ratio), negative LR
Performance of WHO simplified score for eligible antiviral treatment | at 1st OPD visit through initiation of antivirus or 1 year (if not indication for antivirus)
  Gold standard: Eligible antiviral treatment according to EASL criteria Description: performance was define by sensitivity(%), specificity(%), PPV(%), NPV(%), positive LR, negative LR
Performance of REACH-B score for eligible antiviral treatment | at 1st OPD visit through initiation of antivirus or 1 year (if not indication for antivirus)
  Gold standard: Eligible antiviral treatment according to EASL criteria Description: performance was define by sensitivity(%), specificity(%), PPV(%), NPV(%), positive LR, negative LR

SECONDARY OUTCOMES:
Performance of TREAT-B score for eligible antiviral treatment | at 1st OPD visit through initiation of antivirus or 1 year (if not indication for antivirus)
  Gold standard: Eligible antiviral treatment according to Thai guideline criteria Description: performance was define by sensitivity(%), specificity(%), PPV(%), NPV(%), positive LR, negative LR
Performance of WHO simplified score for eligible antiviral treatment | at 1st OPD visit through initiation of antivirus or 1 year (if not indication for antivirus)
  Gold standard: Eligible antiviral treatment according to Thai guideline criteria Description: performance was define by sensitivity(%), specificity(%), PPV(%), NPV(%), positive LR, negative LR
Performance of REACH-B score for eligible antiviral treatment | at 1st OPD visit through initiation of antivirus or 1 year (if not indication for antivirus)
  Gold standard: Eligible antiviral treatment according to Thai guideline criteria Description: performance was define by sensitivity(%), specificity(%), PPV(%), NPV(%), positive LR, negative LR

CONTACTS AND LOCATIONS:
Overall Officials: Watcharasak Chotiyaputta, Assoc prof, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No